CLINICAL TRIAL: NCT02635490
Title: Is Prophylactic Antibiotics Necessary In Otherwise Healthy Adult Patients Undergoing Ureteroscopic Procedures for Ureteral Stones?
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Cheng-Hsing Hsieh, Director,Department of Urology, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 01-X20-068
Record Dates: First submitted 2014-08-06; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Ureteral Stones
Keywords: prophylactic antibiotics, urinary tract infection.
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prophylactic antibiotics

SUMMARY:
The present study aims to investigate the relative efficacy, safety and risk of a single-dose prophylaxis in otherwise healthy adult patients undergoing ureteroscopic procedures for ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

* 100 otherwise healthy adult patients.
* Aged from 20 to 65 years.
* Undergoing ureteroscopic procedures for ureteral stones.

Exclusion Criteria:

* Have the urine road the infection before the surgical operation, the surgical operation once took antibiotics the first 2 week.
* Pregnant or the women been breast feeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort study
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite urinary tract infection confirmed by urinary analysis or urinary culture. | within the first 10 days (plus or minus 5 days) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng-Hsing Hsieh, Taipei, Xindian, Taiwan